CLINICAL TRIAL: NCT03962673
Title: Intestinal Microbiota Changes After Ultra Violet Radiation B Exposure
Brief Title: UVB: Skin to Gut Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Bruce Vallance, Principle Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H17-00303
Record Dates: First submitted 2019-05-22; First posted 2019-05-24 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Healthy
Keywords: Phototherapy; Microbiome; Vitamin D

STUDY DESIGN:
Intervention Model Description: All participants are receiving the same treatment of which the UVB dose is adjusted for the participants Fitzpatrick skin type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UVB- exposure (Experimental): Each participant will receive a pre-determined dose of UVB light. Serum Vitamin D and microbiome samples of each participant will be compared before and after the UVB light exposures.
  Interventions: Radiation: NB-UVB light exposure

INTERVENTIONS:
Radiation: NB-UVB light exposure — Participants are exposed to three low dose Narrow Band UVB light.

SUMMARY:
This research will explore the potential effects of Narrow-Band Ultra Violet B (NB-UVB) radiation on the intestinal microbiota composition and confirm a regulatory skin-to-gut axis during baseline conditions. Changes in the intestinal microbiota composition caused by NB-UVB phototherapy could be beneficial for patients with chronic/auto-inflammatory diseases like inflammatory bowel disease (IBD) by removing dangerous bacteria, increasing beneficial bacteria, and ultimately modulating immune responses.

DETAILED DESCRIPTION:
Purpose:

To explore the potential effects of Narrow-Band Ultra Violet B (NB-UVB) radiation on the intestinal microbiota composition in humans and confirm a regulatory skin-to-gut axis during baseline conditions.

Hypothesis:

Humans exposed to UVB-NB light will show changes in the intestinal microbiota composition with the selection of certain phyla of bacteria.

Justification:

To date, there is no data that describes a biological response to UVB light in the body that affects the intestinal microbiota. Changes in the intestinal microbiota composition caused by NB-UVB phototherapy could be beneficial for patients with chronic/auto-inflammatory diseases like IBD by removing dangerous bacteria, increasing beneficial bacteria, and ultimately modulating immune responses.

Objectives:

1. Establish if there is a skin regulatory response towards NB-UVB light in humans.
2. Examine what changes in the microbiota composition can be observed on bacterial phyla and class level.
3. Determine if this research is worth pursuing in a larger cohort.

Research design:

During the first visit, the skin type will be assessed by using the Fitzpatrick skin type questionnaire.

Subsequently, subjects will be exposed three times within one week to full body NB-UVB light in The Skin Care Centre to a sub erythemic dose (cause slight redness of the skin but not burning). The exposures will happen during the winter months to prevent UVB exposure from the sun during daily activities to interfere with our observations. Stool samples will be collected before the first exposure (2x) and after the last exposure (2x) to analyze the microbiota composition. Also, serum vitamin D (25-hydroxy vitamin D) will be measured before and after the UVB exposure as a marker of previous UVB exposure before the experiment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian females
* Fitzpatrick skin type I, II or III

Exclusion Criteria:

* Skin photosensitivity due to medication
* Been on vacation to a sunny destination three months before enrollment
* Visit tanning beds on a regular basis in the past

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy Caucasian females
Enrollment: 23 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
Serum vitamin D | 1 week
  The effect of UVB light exposures on the serum vitamin D concentrations
Microbiome | Before and after the UVB exposures (1 week apart)
  Changes in the fecal microbiome composition after the UVB light exposures

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A. Vallance, PhD, Principal Investigator — BC Childrens Hospital Research Institute
Locations (1):
- BC Childrens Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Participant information remains deidentified.

REFERENCES:
- [Derived] Bosman ES, Albert AY, Lui H, Dutz JP, Vallance BA. Skin Exposure to Narrow Band Ultraviolet (UVB) Light Modulates the Human Intestinal Microbiome. Front Microbiol. 2019 Oct 24;10:2410. doi: 10.3389/fmicb.2019.02410. eCollection 2019. PMID 31708890

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/73/NCT03962673/Prot_SAP_000.pdf